CLINICAL TRIAL: NCT02834559
Title: Prophylactic Intravitreal 5-Fluorouracil and Heparin to Prevent PVR in High-risk Patients With Retinal Detachment.
Acronym: PRIVENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitätsklinikum Köln (Other)
Collaborators: German Research Foundation (Other); The Clinical Trials Centre Cologne (Other); Pharmacy of the University Hospital Erlangen (Unknown); Institute of Medical Statistics, Informatics and Epidemiology (IMSIE) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: uni-koeln-1782; 2015-004731-12 (EudraCT Number)
Record Dates: First submitted 2016-07-12; First posted 2016-07-15 (Estimated); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Rhegmatogenous Retinal Detachment; High-risk for Proliferative Vitreoretinopathy (PVR)
MeSH Terms: interventions — Fluorouracil; Heparin, Low-Molecular-Weight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adjuvant therapy with 5-FU and LMWH (Active Comparator): Intraoperative adjuvant application of 5-fluorouracil (5-FU) and low molecular weight heparin (LMWH) via intraocular infusion during routine pars plana vitrectomy (PPV) in high-risk patients for proliferative vitreoretinopathy (PVR) with primary rhegmatogenous retinal detachment (RRD).
  Interventions: Drug: 5-fluorouracil and low molecular weight heparin
- Standard of care (Placebo Comparator): Routinely used intraocular infusion with balanced salt solution (BSS) during routine pars plana vitrectomy (PPV) in high-risk patients for proliferative vitreoretinopathy (PVR) with primary rhegmatogenous retinal detachment (RRD).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 5-fluorouracil and low molecular weight heparin — Intraoperative adjuvant application of 5-fluorouracil (5-FU) and low molecular weight heparin (LMWH) via intraocular infusion during routine pars plana vitrectomy (PPV).
  Arms: Adjuvant therapy with 5-FU and LMWH
Drug: Placebo — Routinely used intraocular infusion with balanced salt solution (BSS) during routine pars plana vitrectomy (PPV).
  Arms: Standard of care

SUMMARY:
This study investigates the effectiveness of a simple treatment to prevent proliferative vitreoretinopathy (PVR).

Intraoperative intravitreal 5-fluorouracil (5-FU) and low molecular weight heparin (LMWH) is used as a prophylactic therapy in high-risk patients with primary rhegmatogenous retinal detachment (RRD). Our major motivation is to reduce the incidence of PVR in the group that receives the trial drug.

DETAILED DESCRIPTION:
Proliferative vitreoretinopathy (PVR) is a common cause for postoperative failure after vitreoretinal surgery for primary RRD. There is no standard-therapy to prevent PVR. Several attempts using chemotherapeutic agents have been undertaken to prevent this proliferation-process, but none of these was introduced into routine clinical practice.

Until recently, it has been challenging to identify patients with high risk for postoperative PVR formation. This is especially important, because in this trial treatment with the trial drug will be restricted to patients at high risk for PVR only.

Patients are assigned to the following treatment arms (1:1):

(A) Intraoperative adjuvant application of 5-fluorouracil (5-FU) and low molecular weight heparin (LMWH) via intraocular infusion during routine pars plana vitrectomy (PPV) in high-risk patients for proliferative vitreoretinopathy (PVR) with primary rhegmatogenous retinal detachment (RRD).

Versus:

(B) Routinely used intraocular infusion with balanced salt solution (BSS) during routine PPV.

ELIGIBILITY:
Inclusion Criteria:

1. Primary rhegmatogenous retinal detachment (< 4 weeks) in study eye
2. Scheduled for pars plana vitrectomy for retinal detachment repair without combined cataract surgery in study eye
3. Elevated protein levels in anterior chamber fluid (laser-flare value ≥ 15.0 pc/ms) in study eye
4. Female or male patient ≥ 18 years of age
5. Written informed consent

Exclusion Criteria:

1. Retinal detachment lasting > 4 weeks in study eye
2. Traumatic retinal detachment in study eye
3. Giant retinal tears in study eye (size > 3 clock hours)
4. Visual pre-existing PVR grade C in study eye
5. Retinal dystrophies in study eye
6. Scheduled for combined pars plana vitrectomy and cataract surgery for retinal detachment repair in study eye
7. Chronic inflammatory conditions in study eye
8. Active retinal vascular disease in study eye
9. Proliferative diabetic retinopathy in study eye
10. Manifest uveitis in study eye
11. Endophthalmitis in study eye
12. Perforating and non-perforating trauma in study eye
13. Malignant intraocular tumor in study eye
14. Aphakia in study eye
15. Uncontrolled glaucoma or ocular hypertension in study eye (intraocular pressure ≥ 30 mmHg despite IOP lowering therapy)
16. Previous intraocular surgery except uncomplicated cataract surgery with posterior chamber lens implantation in study eye
17. Cataract surgery in study eye ≤ 3 months ago
18. Previous retinal procedures (laserpexy, cryopexy, intravitreal gas-injection, anti-VEGF or corticosteroid-injection) in study eye ≤ 6 months
19. Other uncontrolled ophthalmologic disorders
20. Single eyed patients (BCVA of fellow eye > 1.0 log MAR, < 0.1 decimal, < 1/10 tenth, or < 6/60 Snellen fraction [m])
21. Evidence or history of alcohol, medication or drug dependency within the last 12 months.
22. Evidence or history (within the last 12 months) of neurotic personality, psychiatric illness that requires or required treatment, epilepsy or suicide risk.
23. Systemic disorders not compatible with adjuvant application of 5-FU and LMWH via intraocular infusion, or not compatible with the local or general anesthesia
24. Any therapy with immunosuppressant or chemotherapy ≤ 3 months and during the trial period
25. Participation in another trial of IMPs or devices parallel to, or less than 3 months before screening, or previous participation in this trial.
26. Known to or suspected of not being able to comply with the protocol.
27. Inability to understand the rationale of this trial or the study aim
28. Any dependency of the patient to the Investigator or the trial site, e.g. employees with direct involvement in the proposed trial or in other trials under the direction of this Investigator or trial site, as well as family members of the employees or the Investigator.
29. Positive urine pregnancy test, pregnancy or breastfeeding mother.
30. Women of child bearing potential without satisfactory contraception, i.e. hormonal contraceptives for at least 14 days before trial enrolment, IUD, double barrier (women of child bearing age must be counselled about the use of adequate contraception).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Proliferative Vitreoretinopathy (PVR) grade CP (posterior - full thickness retinal folds in clock hours) 1 or higher [yes/no] | within 12 weeks

SECONDARY OUTCOMES:
PVR grade CP 1 or higher [yes/no] | within 6 weeks
PVR grade CA (anterior - full thickness retinal folds in clock hours) 1 or higher [yes/no] | within 6 weeks and 12 weeks
Degree of PVR (PVR grade CA 1-12, PVR grade CP 1-12 (in clock hours)) | within 6 weeks and 12 weeks
Best Corrected Visual Acuity (BCVA) measured by ETDRS charts | within 6 weeks and 12 weeks
Retinal reattachment after primary intervention [yes/no] | within 6 weeks and 12 weeks
Number of retinal re-detachments and if present due to PVR [yes/no] | within 6 weeks and 12 weeks
Number and extent of surgical procedures necessary to achieve retinal reattachment | within 12 weeks
Occurrence of at least one drug-related adverse event that affects the study eye [yes/no] | within 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Friederike Schaub, PD. Dr., Principal Investigator — Department of Ophthalmology, University of Cologne
Locations (13):
- Germany (13):
  - Augenklinik Uniklinik Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - STZ eyetrial am Department für Augenheilkunde, Tübingen, Baden-Wurttemberg
  - Klinik und Poliklinik für Augenheilkunde Uniklinik Hamburg Eppendorf, Hamburg, Hamburg
  - Augenklinik Uniklinik Bonn, Bonn, North Rhine-Westphalia
  - Augenklinik der Universität zu Köln, Cologne, North Rhine-Westphalia
  - Universitäts-Augenklinik Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Augenärzte am St. Franziskushospital Münster Augenklinik, Münster, North Rhine-Westphalia
  - Knappschaftskrankenhaus Sulzbach Augenklinik Sulzbach, Sulzbach, Saarbrücken
  - Uniklinik Leipzig Klinik und Poliklinik für Augenheilkunde, Leipzig, Saxony
  - Universitätsaugenklinik Göttingen, Göttingen
  - Universitätsaugenklinik Kiel, Kiel
  - Augenklinik TU München, München
  - Universitätsaugenklinik Regensburg, Regensburg

REFERENCES:
- [Derived] Schaub F, Hoerster R, Schiller P, Felsch M, Kraus D, Zarrouk M, Kirchhof B, Fauser S. Prophylactic intravitreal 5-fluorouracil and heparin to prevent proliferative vitreoretinopathy in high-risk patients with retinal detachment: study protocol for a randomized controlled trial. Trials. 2018 Jul 16;19(1):384. doi: 10.1186/s13063-018-2761-x. PMID 30012187